CLINICAL TRIAL: NCT02401698
Title: Exploring Cerebellar Inhibition of the Motor Cortex in Stroke Patients
Status: Suspended | Type: Observational
Why Stopped: To perform a interim analyzes
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 36990314.4.0000.0068
Record Dates: First submitted 2014-11-26; First posted 2015-03-30 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Stroke
Keywords: Stroke; Transcranial Magnetic Stimulation; Neuronal Plasticity; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Functional clinical and TMS diagnostic — Functional clinical and TMS diagnostic examination to evaluate corticospinal motor tract activity and corticocerebellar tract activity and its relation with stroke recovery

SUMMARY:
The past 10 years of research in post stroke patients have shown certain types of rehabilitation can help neuronal plasticity of the brain. Transcranial magnetic stimulation (TMS) can be used to monitor this plasticity by mapping the brain's function (measuring brain activity). Recent research suggests that TMS can be used for both prognosis (determining future function) and to determine what type of rehabilitation therapy will work best after stroke. The purposes of this research study are to: 1) determine changes in cerebellar activity after motor cortical stroke 2) compare changes in recovery of motor function with changes in cerebellar - motor cortex connections; 3) determine the ability of TMS to "predict" functional outcome after stroke. The primary hypotheses are: 1) functional recovery will be correlated with TMS changes (as measure of motor threshold (MT), intracortical inhibition, cerebellar cerebral inhibition (CBI), motor evoked potentials (MEPs) and recruitment curves; 2) baseline TMS will predict future functional outcomes.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) can be used to monitor this plasticity by mapping the brain's function (measuring brain activity). Recent research suggests that TMS can be used for both prognosis (determining future function) and to determine what type of rehabilitation therapy will work best after stroke. The purposes of this research study are to: 1) determine changes in cerebellar activity after motor cortical stroke 2) compare changes in recovery of motor function with changes in cerebellar - motor cortex connections; 3) determine the ability of TMS to "predict" functional outcome after stroke. The primary hypotheses are: 1) functional recovery will be correlated with TMS changes (as measure of motor threshold (MT), intracortical inhibition, cerebellar cerebral inhibition (CBI), motor evoked potentials (MEPs) and recruitment curves; 2) baseline TMS will predict future functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* one sided ischemic stroke confirmed by radiology
* adults

Exclusion Criteria:

* brainstem stroke
* cerebellar stroke
* seizure with the recent stroke
* any history of uncontrolled seizure
* pregnancy or planning on getting pregnant during the next year
* recent history (past year) of alcohol and drug abuse (due to lack of follow up) Other criteria include TMS exclusions: aneurysm clips, previous surgery over motor cortex, open craniotomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 8 a 19 patients who have suffered a unilateral ischemic stroke up to 2 years and who will undergo motor rehabilitation at the study center will be asked to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Motor function on the Upper Limb Fugl-Meyer Scale and the motor evoked potentials (MEP) on the Transcranial Magnetic Stimulation. | 3 months
  To explore the relationship between the cerebellar brain inhibition - CBI and motor function of upper extremities of patients with stroke. The cerebellar brain inhibition will be assessed by Transcranial Magnetic Stimulation (TMS) and the motor function of the upper extremities by the Upper Limb Fugl-Meyer Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Linamara Rizzo Battistella, MD PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Centro de Pesquisa Clínica do Instituto de Medicina e Reabilitação do HCFMUSP, São Paulo, São Paulo, Brazil